CLINICAL TRIAL: NCT04106947
Title: Transition of Care for Patients With Hirschsprung Disease and Anorectal Malformations
Acronym: NOHARM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Skane University Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Anders Telle Hoel, Clinical Fellow, Oslo University Hospital
Other Study IDs: 18/19101
Record Dates: First submitted 2019-09-20; First posted 2019-09-27 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Anorectal Malformations; Transition; Quality of Life; Hirschsprung Disease
MeSH Terms: conditions — Anorectal Malformations; Hirschsprung Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Hirschsprung and anorectal malformation: Patients with Hirschsprung and anorectal malformation living in Norway
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires

SUMMARY:
Transition from paediatric to adult health care is crucial for preventing deterioration of chronic diseases. At present, transitional care (TC) is not established for patients with the Hirschsprung disease (H) and Anorectal Malformations (ARM). To set up a program for TC and to treat persisting symptoms in adults, data on outcome in adult patients are needed. At present such data are very limited. Therefore, we want to investigate clinical and PROM in H and ARM adolescents and adults. A cross sectional study in all H and ARM patients operated in Norway from 1970-2000 and in all adolescents operated at Oslo University Hospital from 2002-2006 will examine somatic, psychosocial and mental health, and quality of life (QoL). In children operated for H and ARM a large body of evidence shows that bowel problems, reduced QoL and impaired psychosocial and mental health are common. There are papers on sexual and urological impairment in these patients, but large studies on the topic is missing. It is a general assumption among paediatric surgeons that both somatic and mental health problems related to H and ARM improve during adolescence and adult life. Therefore, no standardized guidelines for TC in these patients have been established. Interestingly, very few studies have actually examined H and ARM patients beyond adolescence. Reports from patient organizations showing significant long-term sequels and inadequate understanding of the unique problems of H and ARM patients among health professionals treating adults. Hypothesis:H and ARM adults and adolescents have bowel, urinary and sexual difficulties and reduced QoL, psychosocial and mental health. H and ARM adults receive insufficient treatment of their chronic congenital disease. H and ARM patients with syndromes have particularly bad functional outcome. Anal dilatations and repeated rectal enemas have a negative impact on adolescent psychosocial and mental health. Main aim: Acquire knowledge about long-term bowel, urinary and sexual function, QoL and psychosocial and mental health in adult and adolescent H and ARM patients. Results: from this large study of H and ARM patients will have significant influence on treatment and follow-up, both nationally and internationally. Since very few countries except the Nordic countries have the possibility to follow patients with congenital malformations into adulthood, it is important that studies like this are done.

ELIGIBILITY:
Inclusion Criteria:

Alle patients with Hirschsprung and anorectal malformation

Exclusion Criteria:

None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alle patients with Hirschsprung and anorectal malformations living in Norway
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
questionnaire: BFS | 2 years
  Acquire knowledge about long-term bowel function in adult and adolescent H and ARM patients
questionnaire: DAN-PSS | 2 years
  Acquire knowledge about urinary function in adult and adolescent H and ARM patients
urinary flow-residual | 2 years
  Acquire knowledge about urinary function in adult and adolescent H and ARM patients
questionnaire: PIQS12 and IIEF-5 | 2 years
  Acquire knowledge about sexual function in adult and adolescent H and ARM patients
questionnaire | 2 years
  Acquire knowledge about quality of life in adult and adolescent H and ARM patients
questionnaires | 2 years
  Acquire knowledge about mental Health in adult and adolescent H and ARM patients

SECONDARY OUTCOMES:
Focus Group interviews With adult Hirschsprung's disease (HD) and anorectal malformations (ARM) patients | 2 years
  Acquire knowledge about how adult H and ARM patients have experienced and would design transition from paediatric to adult health care
Questionnaires (impact of event scale) to adolescent and parent. Focus Group interviews will be applied for parents. | 2 years
  Acquire knowledge about the influence of anal dilatations and regular rectal enemas on psychosocial and mental health in adolescents
Focus Group interviews will be applied for parents. | 2 years
  Acquire knowledge about the influence of anal dilatations and regular rectal enemas on psychosocial and mental health in adolescents
Questionnaires to next of kin to syndromic patients | 2 years
  Acquire knowledge about bowel function in adult syndromic H and ARM patients

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bjørnland, Prof, Study Chair — Oslo University Hospital and University of Oslo
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No